CLINICAL TRIAL: NCT01296893
Title: Can Exercise Improve Cancer Associated Cognitive Dysfunction?
Acronym: chemobrain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H10-02774
Record Dates: First submitted 2011-02-09; First posted 2011-02-16 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed exercise control (No Intervention): Participants asked to maintain usual lifestyle and provided with abbreviated version of intervention upon completion of end of study testing.
- Exercise (Experimental): Aerobic exercise Intervention as per below
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 150 minutes/week of aerobic exercise at 60-70% of heart rate reserve (individualized based on baseline VO2 peak test). The intervention is 24 weeks with an exercise progression to reach the full exercise prescription by week 8. Participants are required to attend two 45 minute supervised sessions per week and complete two additional 30 minute sessions independently at home.
  Arms: Exercise

SUMMARY:
Following chemotherapy, some breast cancer survivors report alterations in their ability to remember, concentrate, or think, which can have significant emotional, psychological, and economic impact on their lives. Survivors have also reported feeling frustrated by the response of the medical community, who either may not acknowledge their symptoms or have no treatment options to suggest. Exercise may be a promising treatment, as improvements in cognitive function with exercise have been demonstrated in older adults and other clinical populations.

The investigators will recruit women who have completed chemotherapy for breast cancer (within the past 2 years) and report cognitive changes. Women will be randomly assigned to either a 24-week aerobic exercise intervention or delayed exercise control (offered the same exercise program following the study). At the start and end of the study the investigators will measure: i) performance on four standard neuropsychological tests that measure working memory, learning, and problem solving; ii) a questionnaire on cognitive function and its impact on quality of life; iii) functional magnetic resonance imaging (fMRI) during two of the standard neuropsychological tests which provides information on how the brain is working during the tests.

To knowledge of the investigators this is the first study to examine the effect of an exercise intervention on cognitive function in breast cancer survivors. In addition, the use of fMRI imaging is a new way to approach this research question, and may be more sensitive to change than traditional measures of cognitive function.

DETAILED DESCRIPTION:
Objective 1:

Conduct a randomized trial to test the effectiveness of a 24-week aerobic exercise intervention in adult, female breast cancer survivors with self-reported cognitive changes following chemotherapy.

The investigators will test the following hypotheses:

1. A) The exercise intervention will improve performance on neuropsychological tests of specific cognitive domains of executive function, namely i)selective attention and response inhibition, ii)processing speed and mental flexibility, and iii) verbal memory and learning in exercisers (EX; n=15) versus delayed exercise controls (CON; n=15).

   B) The exercise intervention will reduce self-reported cognitive dysfunction and its impact of function and quality of life, in EX compared to CON, measured as a decreased score on the Functional Assessment Cancer Therapy-Cognition Scale (FACT-Cog).

   Objective 2:

   Conduct analyses on the effect of the intervention on brain activation patterns using functional magnetic resonance imaging (fMRI).

   The investigators will test the following hypotheses:
2. A) At baseline, brain activation patterns will differ in breast cancer survivors reporting cognitive difficulties following chemotherapy compared to breast cancer survivors who have not received chemotherapy (who serve as breast cancer/no chemotherapy controls; not enrolled in the exercise intervention) during neuropsychological tests completed in the scanner.

B) The exercise intervention will result in a decrease in regions of cortical activation, particularly in regions that show higher activation in breast cancer survivors following chemotherapy, compared with no change in controls.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Completed chemotherapy within past 2 years

  * completed for at least 3 months
* Self report cognitive dysfunction following chemotherapy
* Stage I-IIIA breast cancer
* Physically able to undertake moderate to vigorous physical activity program

Exclusion Criteria:

* Self report > 90min/week of moderate physical activity (last 6 months)
* Mini-mental status exam score < 23
* Co-morbid conditions that may alter cognitive testing results (i.e., a clinically diagnosed major depression, anxiety disorder, or other psychiatric condition, meeting DSM IV criteria)
* History of substance abuse
* Other neurological disorder (i.e., head injury, epilepsy, tumour, neurodegenerative disease)
* Ruled ineligible for MRI scanning (i.e., metal implants)

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Stroop Test | Change from baseline at 6 months
  Tests response inhibition, measure number of correct vs incorrect responses

SECONDARY OUTCOMES:
FACT-Cog | Change from baseline at 6 months
  Self-reported cognitive function and quality of life
fMRI analyses | Change from baseline at 6 months
  regions of interest analysis, whole brain patterns of change
Graded exercise test | Change from baseline at 6 months
Hopkins Verbal Learning Test | Change from baseline at 6 months
  Verbal Learning, measure number of recalled and recognized words
Trail Making A & B | Change from baseline at 6 months
  Visual Conceptual and Visuomotor Tracking, measure time taken to complete

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Campbell, PT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Campbell KL, Kam JWY, Neil-Sztramko SE, Liu Ambrose T, Handy TC, Lim HJ, Hayden S, Hsu L, Kirkham AA, Gotay CC, McKenzie DC, Boyd LA. Effect of aerobic exercise on cancer-associated cognitive impairment: A proof-of-concept RCT. Psychooncology. 2018 Jan;27(1):53-60. doi: 10.1002/pon.4370. Epub 2017 Feb 10. PMID 28075038